CLINICAL TRIAL: NCT04375150
Title: Study of Advanced Renal Cell Carcinoma Treatment Patterns and Unmet Needs Using Real World Claims and Electronic Medical Record Data.
Brief Title: Master Protocol to Study Treatment Patterns, Medication Adherence, Health and Economic Outcomes and Unmet Needs in RCC
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181232
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Patients with advanced renal cell carcinoma (RCC)
  Interventions: Drug: Tyrosine kinase inhibitor (TKI); Drug: Immuno-oncology (IO)

INTERVENTIONS:
Drug: Tyrosine kinase inhibitor (TKI) — TKIs
Drug: Immuno-oncology (IO) — IOs

SUMMARY:
The study aims to assess treatment patterns and outcomes in advanced RCC patients in real world clinical practices across various real world databases. Four databases will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older in the year of the index first line therapy prescription.

  * 2 or more RCC diagnoses (ICD-9: 189.0; ICD-10: C64.1, C64.2, C64.9) at least 30 days apart, in the 1 year prior to the index date until 30 days post index date.
  * 2 or more code for secondary malignancy codes indicating possible diagnoses for metastatic disease at least 30 days apart, in the 1 year prior to the index date until 30 days post index date. (ICD-9: xx-199.xx; ICD-10: C77-C79, except ICD9: 198.0 Secondary malignant neoplasm of the kidney and ICD10: C79.0 Secondary malignant neoplasm of the kidney and renal pelvis.)
  * Exploratory sensitivity analyses were performed to review patients with 1 or more diagnosis codes for advanced or metastatic RCC 12 months prior to the index date and 1 or more secondary malignancy codes around the RCC diagnosis dates.
  * Continuous enrollment from 12 months prior to the index date. Patients will be required to have continuous enrollment from their index date until the end of the available data. This will allow for sub-analysis of cohorts with 3 months, 6 months and 12 months of available data

Exclusion Criteria:

* Received advanced treatment prior to the study index date.

  * Prescription records with negative days of supply will be excluded from all the analyses except in cost variable calculation. The day of supply for claims with missing or 0 days will be imputed.
  * Only one RCC diagnosis in the 12 months prior or one mont post index date.
  * Patients with data for analysis (< 3 months post index date)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with RCC
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer INC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with advanced/metastatic renal cell carcinoma (RCC) who initiated treatment for aRCC between 1-Apr-2018 and 31-Jul-2022 were observed. Data was collected retrospectively from various real world claims databases (Truven, Optum, Pharmetrics and the PanTher). Index date was the date of initiation of the aRCC treatment. Data was collected and observed for approximately 35 months (02 December 2019 to 28 October 2022) of this study.
Pre-assignment Details: A total of 355 participants were included in the study.
Groups:
- Axitinib + Pembrolizumab: Participants diagnosed with aRCC who initiated treatment with axitinib + pembrolizumab between 1-Apr-2018 and 31-Jul-2022 were included and observed retrospectively in this study.
- Axitinib + Avelumab: Participants diagnosed with aRCC initiated treatment with axitinib + avelumab between 1-Apr-2018 and 31-Jul-2022 were included and observed retrospectively in this study.
Period: Overall Study
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Started | 340 | 15
Completed | 340 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab | Total
Number analyzed (Participants) | 340 | 15 | 355
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.13 (10.93) | 66.87 (10.45) | 64.25 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 3 | 108
  Male | 235 | 12 | 247
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 1 | 25
  Not Hispanic or Latino | 237 | 8 | 245
  Unknown or Not Reported | 79 | 6 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 0 | 19
  White | 228 | 11 | 239
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 90 | 4 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Line Treatment Regimen
Description: Number of participants with first line treatment regimen prescribed following a primary and secondary diagnosis of advanced/metastatic disease is reported in this outcome measure. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: At index (anytime between 1-Apr-2018 and 31-Jul-2022 [approximately 52 months]); data collected and observed retrospectively over 35 months
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants | 340 | 15

2. Primary Outcome: Number of Participants With Monotherapy and Combination Therapy
Description: Participants who received monotherapy and combination therapy by line of therapy is reported in this outcome measure. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: From the index date until end of enrollment, follow-up or death (maximum of 52 months); data collected and observed retrospectively over 35 months
Population: All eligible participants whose data were retrieved and observed in this study. Here, 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants
  Monotherapy- First Line | 0 | 0
  Monotherapy- Second Line: number analyzed (Participants) | 148 | 8
  Monotherapy- Second Line | 97 | 6
  Monotherapy- Third Line: number analyzed (Participants) | 51 | 3
  Monotherapy- Third Line | 21 | 1
  Monotherapy- Fourth Line: number analyzed (Participants) | 14 | 1
  Monotherapy- Fourth Line | 4 | 1
  Monotherapy- Fifth Line: number analyzed (Participants) | 5 | 1
  Monotherapy- Fifth Line | 5 | 1
  Monotherapy- Sixth Line: number analyzed (Participants) | 1 | 0
  Monotherapy- Sixth Line | 1 |
  Combination therapy- First Line | 340 | 15
  Combination therapy- Second Line: number analyzed (Participants) | 148 | 8
  Combination therapy- Second Line | 51 | 2
  Combination therapy- Third Line: number analyzed (Participants) | 51 | 3
  Combination therapy- Third Line | 30 | 2
  Combination therapy- Fourth Line: number analyzed (Participants) | 14 | 1
  Combination therapy- Fourth Line | 10 | 0
  Combination therapy- Fifth Line: number analyzed (Participants) | 5 | 1
  Combination therapy- Fifth Line | 0 | 0
  Combination therapy- Sixth Line: number analyzed (Participants) | 1 | 0
  Combination therapy- Sixth Line | 0 |

3. Primary Outcome: Time to First Line Therapy
Description: Time to first line therapy was defined as length of time (days) from the first RCC diagnosis to first line therapy prescription. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: From RCC diagnosis to index date (approximately 52 months); data collected and observed retrospectively over 35 months
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Days | 29.00 [18.00 to 52.00] | 25.00 [20.00 to 56.00]

4. Primary Outcome: Duration of Treatment According to Each Line of Therapy
Description: Duration of treatment as per each line of therapy is reported in this outcome measure. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Days
  First Line Therapy | 11.97 [4.85 to 22.05] | 5.90 [2.80 to 16.27]
  Second Line Therapy: number analyzed (Participants) | 148 | 8
  Second Line Therapy | 5.38 [2.50 to 11.70] | 2.58 [1.32 to 4.03]
  Third Line Therapy: number analyzed (Participants) | 51 | 3
  Third Line Therapy | 4.03 [2.10 to 7.03] | 3.43 [1.27 to 11.33]
  Fourth Line Therapy: number analyzed (Participants) | 14 | 1
  Fourth Line Therapy | 2.75 [1.43 to 6.07] | 3.57 [3.57 to 3.57]
  Fifth Line Therapy: number analyzed (Participants) | 5 | 1
  Fifth Line Therapy | 2.53 [2.37 to 3.93] | 0.90 [0.90 to 0.90]
  Sixth Line Therapy: number analyzed (Participants) | 1 | 0
  Sixth Line Therapy | 4.03 [4.03 to 4.03] |

5. Primary Outcome: Number of Participants With Treatment Continuation
Description: Treatment continuation was considered when there was no more than (>) 30-day gap (i.e., persistent treatment) for the index medication during follow-up period. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants | 21 | 1

6. Primary Outcome: Number of Participants With Treatment Interruption
Description: Treatment Interruption was considered in participants with gaps in treatment greater than allowable gap but who restart the same medication with no indication of switching or augmentation. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants | 171 | 6

7. Primary Outcome: Time to Treatment Interruption
Description: Time from index medication to treatment discontinuation for those within treatment interruptions (>30 day gaps). Represents the time between index and end of last treatment, including any treatment gaps. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study. Here, 'Overall Number of Participants Analyzed' signified participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 171 | 6
Months | 2.10 [0.70 to 4.20] | 1.05 [0.43 to 2.55]

8. Primary Outcome: Number of Participants With Treatment Switch or Augmentation
Description: Number of participants who had treatment switch or augmentation were reported in this outcome measure. Augmentation was defined as addition of treatment to initial therapy prescribed, i.e, initiation of a new therapy different from the initial therapy while continuation of the initial therapy. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants
  Treatment Switch | 146 | 8
  Treatment Augmentation | 2 | 0

9. Primary Outcome: Number of Participants According to Lines of Therapy
Description: Number of participants as per the lines of treatment were reported in this outcome measure. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants
  First Line Therapy | 340 | 15
  Second Line Therapy | 148 | 8
  Third Line Therapy | 51 | 3
  Fourth Line Therapy | 14 | 1
  Fifth Line Therapy | 5 | 1
  Sixth Line Therapy | 1 | 0

10. Primary Outcome: Number of Participants According to Sequence of Therapies for Metastatic Renal Cell Carcinoma (mRCC)
Description: Number of participants according to the sequence of therapies received for mRCC were reported in this outcome measure. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants
  Avelumab,Axitinib | 0 | 7
  Avelumab, Axitinib/ Axitinib, Pembrolizumab | 0 | 1
  Avelumab, Axitinib/ Cabozantinib | 0 | 1
  Avelumab,Axitinib/ Cabozantinib/ Cabozantinib, Nivolumab/ Tivozanib/ Pazopanib | 0 | 1
  Avelumab,Axitinib/ Cabozantinib/ Everolimus, Lenvatinib | 0 | 1
  Avelumab,Axitinib/ Cabozantinib/ Pazopanib | 0 | 1
  Avelumab, Axitinib/ Ipilimumab, Nivolumab | 0 | 1
  Avelumab, Axitinib/ Nivolumab | 0 | 1
  Avelumab, Axitinib/ Pembrolizumab | 0 | 1
  Axitinib,Pembrolizumab | 192 | 0
  Axitinib,Pembrolizumab/ Axitinib (PEM-AXI), leuprolide, Pembrolizumab | 1 | 0
  AXI,PEM/ AXI,Leuprolide,PEM/ Abiraterone,AXI,PEM/Abiraterone,Axitinib,Leuprolide, PEM | 1 | 0
  AXI, PEM/ AXI, PEM/ Cabozantinib | 1 | 0
  AXI, PEM/ Bevacizumab/ Cabozantinib | 1 | 0
  AXI, PEM/ Bevacizumab- Awwb/ Bevacizumab/ Temsirolimus/ Bevacizumab- Awwb | 1 | 0
  AXI, PEM/ Bevacizumab-Awwb/ Cabozantinib | 1 | 0
  AXI, PEM/ Bevacizumab-Awwb, Everolimus | 1 | 0
  AXI, PEM/ Cabozantinib | 48 | 0
  AXI, PEM/ Cabozantinib/Bevacizumab- Awwb | 1 | 0
  AXI, PEM/ Cabozantinib/Cabozantinib, Nivolumab | 4 | 0
  AXI, PEM/ Cabozantinib/ Cabozantinib, PEM/ Everolimus, Lenvatinib | 1 | 0
  AXI, PEM/ Cabozantinib/ Clinical Study Drug (CSD)/ Everolimus, Lenvatinib/ Belzutifan | 1 | 0
  AXI, PEM/ Cabozantinib/ Everolimus, Lenvatinib | 4 | 0
  AXI, PEM/ Cabozantinib/ Everolimus, Lenvatinib/ Bevacizumab -Bvzr, Erlotinib | 1 | 0
  AXI, PEM/ Cabozantinib/ Everolimus, Lenvatinib/ CSD | 1 | 0
  AXI, PEM/ Cabozantinib/ Everolimus,Lenvatinib/ Ipilimumab, Nivolumab | 1 | 0
  AXI, PEM/ Cabozantinib/ Everolimus, Lenvatinib, Tivozanib | 1 | 0
  AXI, PEM/ Cabozantinib/ Ipilimumab, Nivolumab | 2 | 0
  AXI, PEM/ Cabozantinib/ Ipilimumab, Nivolumab/ Everolimus, Lenvatinib | 1 | 0
  AXI, PEM/ Cabozantinib/ Pazopanib/ Ipilimumab, Nivolumab | 1 | 0
  AXI, PEM/ Cabozantinib/ Pazopanib- Lenvatinib, Pembrolizumab/ Tivozanib | 1 | 0
  AXI, PEM/ Cabozantinib/Tivozanib/ Ipilimumab, Nivolumab | 1 | 0
  AXI, PEM/ Cabozantinib,CSD | 1 | 0
  AXI, PEM/ Cabozantinib,Nivolumab | 6 | 0
  AXI, PEM/ Cabozantinib,Nivolumab/ Everolimus,Lenvatinib | 1 | 0
  AXI, PEM/ Cabozantinib,Nivolumab,PEM/ Everolimus,Lenvatinib | 1 | 0
  AXI, PEM/ Cabozantinib,PEM | 6 | 0
  AXI, PEM/Chlorambucil,Obinutuzumab/ Rituximab | 1 | 0
  AXI, PEM/ CSD | 2 | 0
  AXI, PEM/ CSD/ Cabozantinib | 1 | 0
  AXI,PEM/ CSD,Cyclophosphamide,Daratumumab/Hyaluronidase- Fihj,Fludarabine/ Cabozantinib,Nivolumab | 1 | 0
  AXI, PEM/ CSD,Cyclophosphamide,Fludarabine/ Cabozantinib,Nivolumab | 1 | 0
  Axitinib,Pembrolizumab/CSD,Gemcitabine | 1 | 0
  AXI, PEM-Doxorubicin,PEM/ Cabozantinib | 1 | 0
  AXI, PEM/ Everolimus | 1 | 0
  AXI, PEM/ Everolimus/ Pazopanib | 1 | 0
  AXI, PEM/ Everolimus,Lenvatinib | 5 | 0
  AXI, PEM/ Everolimus,Lenvatinib/ Cabozantinib/ Everolimus | 1 | 0
  AXI, PEM/ Everolimus,Lenvatinib/ Cabozantinib,Nivolumab | 1 | 0
  AXI, PEM/ Everolimus,Lenvatinib/ Ipilimumab,Nivolumab | 1 | 0
  AXI, PEM/ Everolimus,Lenvatinib,Pembrolizumab | 1 | 0
  AXI, PEM/ Gemcitabine,Paclitaxel Protein-Bound,Pembrolizumab | 1 | 0
  AXI, PEM/ Hydroxyurea,Pembrolizumab | 1 | 0
  AXI, PEM/ Ipilimumab,Nivolumab | 9 | 0
  AXI, PEM/ Ipilimumab,Nivolumab/ Cabozantinib | 2 | 0
  AXI, PEM/ Ipilimumab,Nivolumab/ Cabozantinib,Ipilimumab,Nivolumab | 1 | 0
  Axitinib,Pembrolizumab/ Ipilimumab,Nivolumab/ CSD | 1 | 0
  AXI, PEM/ Ipilimumab,Nivolumab/ Everolimus,Lenvatinib | 1 | 0
  AXI, PEM/ Lenvatinib | 2 | 0
  AXI, PEM/ Lenvatinib, Pembrolizumab | 1 | 0
  AXI, PEM/ Leuprolide/ Bicalutamide,Leuprolide | 1 | 0
  AXI, PEM/ Nivolumab/ Cabozantinib | 2 | 0
  AXI, PEM/ Nivolumab/ Cabozantinib,Nivolumab | 1 | 0
  AXI, PEM/ Pazopanib | 2 | 0
  AXI, PEM/ Pazopanib/ Cabozantinib/ Everolimus,Lenvatinib/ Sunitinib/ Tivozanib | 1 | 0
  AXI, PEM/ Pazopanib/ Cabozantinib,Nivolumab | 1 | 0
  AXI, PEM/ Pazopanib/ Everolimus,Lenvatinib | 1 | 0
  AXI, PEM/ PEM | 7 | 0
  AXI, PEM/ PEM,Sunitinib | 1 | 0
  AXI, PEM/ Sunitinib/ Pembrolizumab,Sunitinib | 1 | 0
  AXI, PEM/ Sunitinib/Tivozanib/ Cabozantinib/ Tivozanib | 1 | 0

11. Primary Outcome: Number of Participants According to Their Status at End of Follow-up
Description: Number of participants according to their status (death, end of enrollment and end of data availability) at end of follow-up were observed and included in this outcome measure. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: At end of enrollment, follow-up or death (maximum of 52 months) (data collected and observed retrospectively over 35 months)
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Participants
  Death | 161 | 11
  End of enrollment | 104 | 2
  End of data availability | 75 | 2

12. Primary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from first-line therapy start to treatment discontinuation for any reason, including switched, augmented therapy, end of enrollment or death. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Months | 2.57 [2.10 to 2.90] | 1.83 [0.93 to 4.37]

13. Primary Outcome: Percentage of Participants With Treatment Discontinuation
Description: Percentage of participants with treatment discontinuation was defined as the percentage of participants with gap in therapy greater than 30 days and who did not begin a new treatment. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Percentage of participants | 80 | 80

14. Primary Outcome: Percentage of Participants Alive at 3 Months
Description: Percentage of participants who were alive at 3 months is reported in this outcome measure.
Time Frame: At 3 months (data collected and observed retrospectively over 35 months)
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Percentage of participants | 90.29 | 86.67

15. Primary Outcome: Percentage of Participants Alive at 6 Months
Description: Percentage of participants who were alive at 6 months is reported in this outcome measure.
Time Frame: At 3 months (data collected and observed retrospectively over 35 months)
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Percentage of participants | 82.35 | 66.67

16. Primary Outcome: Percentage of Participants Alive at 12 Months
Description: Percentage of participants who were alive at 12 months is reported in this outcome measure.
Time Frame: At 3 months (data collected and observed retrospectively over 35 months)
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Percentage of participants | 67.35 | 40.00

17. Primary Outcome: Overall Survival
Description: OS is defined as the length of time from index date to participant's death. Index date was defined as the date of initiation of the aRCC treatment.
Time Frame: as for outcome 2
Population: All eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
Number analyzed (Participants) | 340 | 15
Days | 29.43 [24.17 to 37.53] | 11.97 [4.83 to 28.47]

ADVERSE EVENTS:
Time Frame: For all-cause mortality: From the index date until end of enrollment, follow-up or death (maximum of 52 months); data collected and observed retrospectively over 35 months. Data for non-serious adverse events and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs.
Description: This observational retrospective study retrieved data from electronic medical records and claims and the data existed as structured data or combination of existing structured and unstructured data. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event could not be met, hence safety data were not collected and reported.
Arm/Group | Axitinib + Pembrolizumab | Axitinib + Avelumab
All-Cause Mortality (participants affected / at risk) | 161/340 | 11/15
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04375150/Prot_SAP_000.pdf